CLINICAL TRIAL: NCT07046871
Title: Effectiveness of an Adapted Basketball Program With and Without Video Support in Adolescents With Obesity: A Randomized Controlled Trial
Brief Title: Effectiveness of Adapted Basketball Programs in Adolescents With Obesity (ABBA)
Acronym: ABBA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sfax (Other)
Responsible Party: Principal Investigator, Antonella Muscella, Associate Professor of Sport Sciences, University of Salento, University of Salento
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 048/2022; 048/2022 (Other: Ethics Committee of the Faculty of Medicine of Sfax)
Record Dates: First submitted 2025-06-05; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Obesity
Keywords: Obesity, Adolescents, Physical Activity, Basketball Intervention, Adapted Physical Education, Motivation, Physical Fitness, Randomized Controlled Trial
MeSH Terms: conditions — Obesity; Motor Activity | interventions — Adiposity

STUDY DESIGN:
Intervention Model Description: Three-arm parallel-group randomized controlled trial. Participants were randomly assigned to one of three intervention arms: (i) an adapted basketball program with pre-session video summaries (ADAPT+VID), (ii) an adapted basketball program without video supplementation (ADAPT), or (iii) a traditional basketball program without specific pedagogical modifications (CONT).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Adapted Basketball Program with Video Support (ADAPT+VID) (Experimental): Adapted basketball program without video supplementation.(ADAPT)
  Interventions: Behavioral: 1. Intervention Name (Arm 1) Name: Adapted Basketball Program with Video Support Type: Behavioral Description: A 7-week basketball intervention for adolescents with obesity, combining pedagogically a
- ADAPT (Experimental): Adapted basketball program without video supplementation.
  Interventions: Behavioral: ADAPT Adapted Basketball Program
- CONTROL (No Intervention): Traditional basketball program with no pedagogical modifications.

INTERVENTIONS:
Behavioral: 1. Intervention Name (Arm 1) Name: Adapted Basketball Program with Video Support Type: Behavioral Description: A 7-week basketball intervention for adolescents with obesity, combining pedagogically a — A 7-week basketball intervention for adolescents with obesity, combining pedagogically adapted activities with pre-session video instruction delivered via a private Facebook group.
  Other Names: Adapted Basketball Program with Video Support (ADAPT+VID)
  Arms: Adapted Basketball Program with Video Support (ADAPT+VID)
Behavioral: ADAPT Adapted Basketball Program — A 7-week adapted basketball intervention including non-competitive, inclusive drills tailored to adolescents with obesity, without any video supplementation.
  Other Names: Adapted Basketball Program
  Arms: ADAPT

SUMMARY:
This study aims to evaluate the effects of different basketball training programs on adolescents with obesity. The objective is to assess how these programs influence body weight, physical fitness, motivation to exercise, and basketball skills.

Three types of programs are being compared:

* A specially adapted basketball program with pre-session instructional video lessons.
* The same adapted program without video supplementation.
* A regular basketball program without pedagogical modifications.

Participants are adolescents aged 15 to 17 years with moderate obesity who will engage in one of the programs for seven weeks, with one training session per week.

Body weight, physical fitness, motivation, and basketball skills will be measured before and after the intervention to determine which approach is most effective.

The study aims to identify engaging and effective methods for promoting physical activity, health, and basketball skill development in adolescents with obesity.

DETAILED DESCRIPTION:
This randomized controlled trial (RCT) includes three parallel intervention arms designed to evaluate the effects of different basketball teaching programs on adolescents with obesity. The intervention spans seven consecutive weeks and consists of one structured basketball session per week, each lasting 60 minutes and delivered during regular physical education (PE) classes.

A total of 55 adolescents (33 females and 22 males), aged 15 to 17 years and classified as having moderate obesity (BMI: 30-34.9 kg/m²), were recruited from a secondary school in the Sidi Bouzid region of Tunisia. Participants were randomly assigned using a computer-generated sequence to one of the following groups:

* ADAPT+VID Group (n = 19): An adapted basketball program enriched with pre-session instructional video summaries.
* ADAPT Group (n = 18): The same adapted basketball program without video supplementation.
* CONT Group (n = 18): A traditional basketball program without pedagogical modifications.

Pre- (T0) and post-intervention (T1) assessments included: (i) anthropometric measurements (BMI), (ii) physical fitness tests, (iii) evaluations of technical basketball performance (passing, dribbling, shooting), and (iv) assessments of motivation. Motivation was assessed following the first and final sessions.

Each session was structured into three phases: a standardized warm-up (15 minutes), a main instructional phase (40 minutes), and a cool-down period (5 minutes). The adapted program was tailored to the specific needs of adolescents with obesity by modifying drills, reducing competitiveness, and incorporating extended recovery and instructional periods. Pre-session videos in the ADAPT+VID group were uploaded to a private Facebook group 48 hours prior to each session and engagement was monitored.

The study received approval from the appropriate institutional ethics committee and was conducted in accordance with the Declaration of Helsinki. Written informed consent was obtained from all participants and their legal guardians prior to enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 15 and 17 years
* Body mass index (BMI) within the moderate obesity range (30-34.9 kg/m²)
* No history of musculoskeletal, neurological, or orthopedic disorders that could impair physical performance in the six months preceding the study
* Normal or corrected-to-normal vision
* Regular attendance in physical education (PE) classes

Exclusion Criteria:•

* History of musculoskeletal, neurological, or orthopedic disorders that could impair physical performance in the six months preceding the study
* Visual impairments not corrected to normal vision
* Irregular attendance or absence from physical education (PE) classes

Ages: 15 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Change in Body Mass Index (BMI) in kg/m² | From baseline (pre-intervention) to after 7 weeks of intervention
  Body Mass Index (BMI) will be calculated using the formula: weight (kg) / height (m²). Weight will be measured using a calibrated digital scale and height using a wall-mounted stadiometer. BMI will be assessed at baseline and after 7 weeks to evaluate the effects of the basketball training intervention on body composition in adolescents with moderate obesity.

SECONDARY OUTCOMES:
Change in Cardiorespiratory Fitness Assessed by Intermittent Fitness Test 15-15. -Unit of Measure: Meters (total distance covered)(Spartacus Test). -Unit of Measure: Meters (total distance covered) | Baseline (pre-intervention)and after 7 weeks
  Cardiorespiratory fitness will be assessed using the 15-15 intermittent fitness test (Spartacus Test), a shuttle run test designed for overweight and obese adolescents. The test involves 15-second running intervals alternated with 15-second passive recovery over a 40-meter distance, with progressive speed increases starting at 5 km/h and increasing by 0.5 km/h per stage. The test concludes when the participant fails to maintain pace for two consecutive intervals or stops due to fatigue. The total distance covered will be used to estimate cardiorespiratory fitness (VO₂peak). The Spartacus test is validated for this population and demonstrates high test-retest reliability (ICC > 0.90).
Change in Situational Motivation (SIMS) Scores. - Unit of Measure: Units on the Situational Motivation Scale (SIMS), a 7-point Likert scale with minimum score 1 and maximum score 7. | Baseline (Session 1) and post-intervention (Session 7, 7 weeks after baseline)
  Motivation was assessed using the Situational Motivation Scale (SIMS), a validated 16-item questionnaire evaluating four subdimensions: intrinsic motivation, identified regulation, external regulation, and amotivation. Each item is rated on a 7-point Likert scale (1 = "does not correspond at all" to 7 = "corresponds exactly"). The average score for each subscale was calculated by averaging the corresponding four items (e.g., intrinsic motivation: items 1, 5, 9, 13). Higher scores indicate greater intensity of the respective motivation type.

OTHER OUTCOMES:
Change in Passing Accuracy in Basketball. -Unit of Measure: Points (maximum possible score based on protocol) | From baseline to after 7 weeks of intervention
  Passing accuracy was evaluated using the AAHPERD Passing Test, which requires participants to perform chest passes at six wall targets within 30 seconds. Points are awarded based on precision and rule compliance. The total score is the sum of two scored trials, after one practice attempt. This test has demonstrated strong reliability (r = 0.84-0.97).
Change in Shooting Accuracy in Basketball -Unit of Measure: Points (0 to 50 maximum) | Baseline and after 7 weeks
  Shooting accuracy was assessed using a standardized 10-shot free-throw test from the 4.57-meter line, using FIBA-approved size 6 basketballs. Each shot was scored using a 6-level scale (0-5 points), considering precision and shot quality. Total score was calculated by summing the scores of the 10 attempts.
Change in Dribbling Performance in Basketball. -Unit of Measure: Seconds | Baseline and after 7 weeks
  Dribbling proficiency was evaluated using a timed zigzag cone course (5 cones, 2 meters apart). Participants completed a round-trip dribbling trial; the best of two attempts was retained. Performance was measured in seconds using a stopwatch accurate to 0.01 seconds.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Sfax, Sfax, Tunisia

IPD SHARING:
Plan to Share IPD: No
At this time, there is no plan to share IPD due to limitations in data-sharing infrastructure and ethical considerations. However, de-identified data may be made available in the future upon reasonable request, pending ethical committee approval.

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2024-12-16): https://cdn.clinicaltrials.gov/large-docs/71/NCT07046871/Prot_ICF_000.pdf